CLINICAL TRIAL: NCT05247853
Title: Long-Term Human Papillomavirus Vaccination Effectiveness and Immunity in Rwandan Women Living With and Without Human Immunodeficiency Virus
Brief Title: HPV Vaccine Effectiveness Study in Rwandan Women Living With HIV
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rwanda Military Hospital (Other); University of Rwanda (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-13087; 1U54CA254568-01 (NIH)
Record Dates: First submitted 2022-01-13; First posted 2022-02-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Cervical Cancer; Human Papilloma Virus; Human Immunodeficiency Virus; HPV-Related Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome | interventions — Blood Specimen Collection; Proctoscopy; Colposcopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — De-identified pictures of participants' cervix, blood collection, oral swab specimen, cervical swab specimen and anal swab specimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: HPV-vaccinated women living with HIV
  Interventions: Procedure: Blood collection; Procedure: Oral, cervicovaginal and anal specimen collection; Procedure: Anoscopy & Biopsy of Acetowhite Lesions; Procedure: Colposcopy & Biopsy of Acetowhite Lesions; Procedure: Ablative Treatment; Procedure: LEEP (Loop Electrosurgical Excision Procedure)
- Group 2: HPV-unvaccinated women living with HIV
  Interventions: Procedure: Blood collection; Procedure: Oral, cervicovaginal and anal specimen collection; Procedure: Anoscopy & Biopsy of Acetowhite Lesions; Procedure: Colposcopy & Biopsy of Acetowhite Lesions; Procedure: Ablative Treatment; Procedure: LEEP (Loop Electrosurgical Excision Procedure)
- Group 3: HIV[-] women who are HPV-vaccinated
  Interventions: Procedure: Blood collection; Procedure: Oral, cervicovaginal and anal specimen collection; Procedure: Colposcopy & Biopsy of Acetowhite Lesions

INTERVENTIONS:
Procedure: Blood collection — Blood collection at enrollment visit
Procedure: Oral, cervicovaginal and anal specimen collection — Oral, cervicovaginal and anal specimen collection at enrollment and follow-up visits
Procedure: Anoscopy & Biopsy of Acetowhite Lesions — Used for management in follow-up visits of persistent anal HPV16/18+ in WLWH
  Groups: Group 1; Group 2
Procedure: Colposcopy & Biopsy of Acetowhite Lesions — Used for management in follow-up visits of persistent type-specific high-risk HPV cervicovaginal HPV
Procedure: Ablative Treatment — Use for management in follow-up visits of persistent cervicovaginal HPV 16/18+ in WLWH, as identified in colposcopy and biopsy
  Groups: Group 1; Group 2
Procedure: LEEP (Loop Electrosurgical Excision Procedure) — Use for management in follow-up visits of persistent cervicovaginal HPV 16/18+ in WLWH, as identified in colposcopy and biopsy that ablation ineligible
  Groups: Group 1; Group 2

SUMMARY:
Our study will assess and measure population effectiveness of prophylactic HPV vaccine in reducing cervical, anal, and/or oral prevalent and 6-month persistent infections among HPV-vaccinated and 757 HPV-unvaccinated Rwandan WLWH aged 18-26 years. Additional objectives include the quantification & examination of long-term antibody (into young adulthood) responses to HPV vaccination and to validate the performance (e.g., sensitivity and specificity) of a low-cost, POC (point-of-care) anti-HPV16 antibody test to determine/confirm HPV vaccination status. The findings for this study will provide necessary evidence regarding the long-term protection afforded by HPV vaccination in WLWH living in SSA, who are at the greatest risk of HPV-related cancers.

DETAILED DESCRIPTION:
Cervical cancer is the 4th most common cancer and cause of cancer-related death in women globally; in many lower-resource settings, especially sub-Saharan Africa (SSA), it is the most common. Virtually all cervical cancer and precancer are caused by 12-15 high-risk human papillomavirus (HPV) types. HPV16 causes approximately 55-60% and HPV18 causes approximately 10-15% of cervical cancer while the remaining 12 HPV types cause the remaining 25-30% of cervical cancer. High-risk HPV, predominately HPV16, also causes most anal, vulvar, vaginal, and penile cancers and a significant proportion of oropharyngeal cancers. Prophylactic HPV vaccines have been developed and have been shown to be nearly 100% protective against incident HPV infection and related abnormalities in the general population. However, the evidence for the effectiveness of prophylactic HPV vaccines in women living with human immunodeficiency virus (HIV) (WLWH) is less clear. HIV infection increases the risk of cervical cancer due to an impaired immune response to HPV.

Rwanda is a high-burden cervical cancer country where the prevalence of HIV is 3.7% among adult women, with higher HIV prevalence among young women (1). In 2011, Rwanda implemented a national HPV vaccination program with Gardasil®, which protects against HPV16 and HPV18, the two HPV types that cause ~70% of cervical cancer, and HPV6 and HPV11, the two types that cause ~90% of anogenital warts (HPV6/11/16/18). Their program has achieved >90% coverage of the target population, primarily girls aged 12 years, annually. The implementation of a highly successful HPV vaccination program and the high prevalence of HIV, in addition to the research and medical capacity that Albert Einstein College of Medicine (Einstein) has helped to build at the Rwanda Military Hospital (RMH) and University of Rwanda (UR), makes Rwanda the ideal locale to study the long-term effects of HPV vaccination in WLWH.

To answer questions about HPV vaccine effectiveness and immunity in Rwandan WLWH, collaborators at Einstein, RMH, and UR will conduct an observational study of WLWH and HIV-negative (HIV[-]) women who did (birth cohorts 1997 and later) and WLWH who did not (birth cohorts before 1997) receive HPV vaccination through the national vaccination program. The investigators will compare cervicovaginal, anal, and oral prevalent and 6-month persistent HPV6/11/16/18 infections in 757 HPV-vaccinated WLWH to those in 757 unvaccinated WLWH and 757 HPV-vaccinated HIV[-] women. The investigators will also compare the HPV immune response in 548 HPV-vaccinated WLWH to 548 HPV-vaccinated HIV[-] women and the impact of switching from 3 doses to 2 doses of Gardasil® in 2015. Finally, the investigators will investigate the risk factors, including the cervicovaginal microbiome, for prevalent and 6-month persistent HPV infection in young WLWH and HIV[-] women. The long-term goal is to establish a cohort of WLWH in whom we can examine the long-term effectiveness of HPV vaccination in WLWH now and in the future. This contribution is significant as it will establish the population effectiveness of HPV vaccination in WLWH living in SSA, the group of women at the highest risk of cervical cancer, for which there is a dearth of evidence. The proposed research is innovative as it leverages and expands the local research and medical capacity in Rwanda to examine one of the critically unanswered questions about HPV vaccine effectiveness in the context of the World Health Organization's (WHO) call for the elimination of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-28 years. The age of inclusion criteria will likely be restricted as age-specific enrollment goals are met.
* Physically and mentally able and willing to participate in the study.
* Willing to provide written and signed or thumb printed, informed consent.
* Known to be living with HIV (i.e., enrolled in a treatment program), or consent to HIV testing to confirm HIV status.

Exclusion Criteria:

* Have positive pregnancy test or report to be pregnant at the time of visit or less than 6 weeks post-partum (will be asked to make an appointment 6 or more weeks post-partum)
* Report to be menstruating at the time of visit (will be asked to make new appointment)
* History of hysterectomy and no longer have a cervix
* History of treatment for cervical abnormalities after cervical screening
* History of cervical cancer
* Report no previous sexual activity
* HIV status is unknown, and date of birth is 12/31/1995 or earlier
* Because this study has age-specific enrollment goals for WLWH and HIV[-] women, once those enrollment goals are met for each study group, the respective cohorts will be closed and other eligible women will be excluded.

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will recruit women attending collaborating clinics and women from the communities surrounding those clinics into three groups: HPV-vaccinated WLWH (Group 1); HPV-unvaccinated WLWH (Group 2); and HIV[-] women who are HPV-vaccinated (Group 3). The number of doses of HPV vaccination received is dictated by introduction of HPV vaccination in Rwanda. In general, most Rwandan women born in 2003 or later will have been vaccinated with two doses of Gardasil®, women born between 1996 and 2002 will have been vaccinated with three doses of Gardasil®, and women born in 1995 or earlier will be unvaccinated. Therefore, we will recruit by age, which will serve as a useful and very good proxy for HPV vaccination status, which otherwise would be difficult to confirm in real time at enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 3127 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Change in vaccine effectiveness of prophylactic HPV vaccine | Baseline and up to 12 months
  To measure population effectiveness of prophylactic HPV vaccine in reducing cervicovaginal, anal, and/or oral prevalent and 6-12 month persistent infections by HPV6/11/16/18
Change in long-term antibody responses to HPV vaccination | Baseline and up to 12 months
  To quantify, and examine the determinants of, long-term antibody (into young adulthood) responses to HPV vaccination

OTHER OUTCOMES:
Change in HPV natural history study at 6 months | Baseline and 6 months
  Conduct a natural history study to investigate determinants, including cervicovaginal microbiome (CVM), of short-term HPV persistence in young WLWH and HIV[-] women living in a SSA setting

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Yotebieng, MD, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Rwanda Military Hospital, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kundrod KA, Jeronimo J, Vetter B, Maza M, Murenzi G, Phoolcharoen N, Castle PE. Toward 70% cervical cancer screening coverage: Technical challenges and opportunities to increase access to human papillomavirus (HPV) testing. PLOS Glob Public Health. 2023 Aug 16;3(8):e0001982. doi: 10.1371/journal.pgph.0001982. eCollection 2023. PMID 37585432
- [Result] Murenzi G, Mungo C. Impact of the human papillomavirus vaccine in low-resource settings. Lancet Glob Health. 2023 Jul;11(7):e997-e998. doi: 10.1016/S2214-109X(23)00203-6. Epub 2023 May 16. No abstract available. PMID 37207682
- [Result] Murangwa A, Desai KT, Gage JC, Murenzi G, Tuyisenge P, Kanyabwisha F, Musafili A, Kubwimana G, Mutesa L, Anastos K, Kim HY, Castle PE. Agreement between Xpert and AmpFire tests for high-risk human papillomavirus among HIV-positive women in Rwanda. Afr J Lab Med. 2022 Oct 19;11(1):1827. doi: 10.4102/ajlm.v11i1.1827. eCollection 2022. PMID 36353194
- [Result] Murenzi G, Shumbusho F, Hansen N, Munyaneza A, Gage JC, Muhoza B, Kanyabwisha F, Pierz A, Tuyisenge P, Anastos K, Castle PE. Long-term human papillomavirus vaccination effectiveness and immunity in Rwandan women living with and without HIV: a study protocol. BMJ Open. 2022 Aug 25;12(8):e061650. doi: 10.1136/bmjopen-2022-061650. PMID 36008069
- [Result] Mukherjee A, Ye Y, Wiener HW, Kuniholm MH, Minkoff H, Michel K, Palefsky J, D'Souza G, Rahangdale L, Butler KR, Kempf MC, Sudenga SL, Aouizerat BE, Ojesina AI, Shrestha S. Variations in Genes Encoding Human Papillomavirus Binding Receptors and Susceptibility to Cervical Precancer. Cancer Epidemiol Biomarkers Prev. 2023 Sep 1;32(9):1190-1197. doi: 10.1158/1055-9965.EPI-23-0300. PMID 37410084

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT05247853/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT05247853/ICF_002.pdf